CLINICAL TRIAL: NCT01943786
Title: Prospective, Non-Interventional Study of K-ras Status Switch in K-ras Native Patients With Metastatic Colorectal Tumors Treated With FOLFIRI-Cetuximab as First-line Treatment
Brief Title: RAS Switch in Patients With Metastatic RAS Native Colorectal Tumors Treated With 1st Line FOLFIRI-Cetuximab
Acronym: BEAMING
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sofia Perea, Director Clinical Trials Unit. (Other)
Responsible Party: Sponsor-Investigator, Sofia Perea, Director Clinical Trials Unit., Director Clinical Research Unit, Grupo Hospital de Madrid
Organization: Grupo Hospital de Madrid (Other)
Other Study IDs: BEAMING
Record Dates: First submitted 2013-04-29; First posted 2013-09-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Wild type KRAS
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FOLFIRI + Cetuximab: Patients with advanced colorectal cancer and wild-type KRAS will receive FOLFIRI + Cetuximab according to regular clinical practice
  Interventions: Drug: FOLFIRI + Cetuximab

INTERVENTIONS:
Drug: FOLFIRI + Cetuximab — Patients will receive study treatment (FOLFIRI + Cetuximab) according to regular clinical practice

SUMMARY:
Adenocarcinoma of the colon and rectum is a common, serious disease and it is the second cause of death from cancer in Spain.

The prognosis of CRC depends to a great extent on its stage when diagnosed. Patients with advanced disease, who present up to 40% of all patients, have a poor prognosis. Although the application of modern chemotherapy and radiotherapy treatments obtains median survival periods of around 24 months, the proportion of patients with advanced disease who obtain a cure is low.

Systemic treatment of advanced CRC has changed considerably in the last ten years with the introduction of active drugs such as oxaliplatin, irinotecan, and capecitabine. The most commonly used first line regimens are 5-Fluorouracil-Leucovorin-Oxaliplatin (FOLFOX), Capecitabine-Oxaliplatin (XELOX), 5-Fluorouracil-Leucovorin-Irinotecan (FOLFIRI) and, to a lesser extent, Capecitabine-Irinotecan (XELIRI). Chemotherapy regimens are combined with different agents against therapeutic targets, three of which are effective in colon cancer: bevacizumab, which targets vascular endothelial growth factor (VEGF) and cetuximab or panitumumab, which target the epidermal growth factor receptor (EGFR).

The use of cetuximab and panitumumab is not recommended in patients with KRAS mutations and the combination of a VEGF and EGFR agents is not beneficial.

Two recent studies results have identified KRAS mutations as frequent drivers of acquired resistance to cetuximab and panitumumab in colorectal cancer patients. The conclusions indicate that the emergence of KRAS mutant clones can be detected non-invasively months before radiographic progression by a DNA Blood Test (Inostics´BEAMing Technology).

Centro Integral Oncológico Clara Campal (CIOCC) is aiming to undertake a pioneer project aimed at integrating the analysis of KRAS switch status by BEAMing Technology in patients with metastatic colorectal cancer, tumor KRAS wild-type and BEAMing wild-type treated with first line FOLFIRI-cetuximab

In naive chemotherapy tumor-KRAS wild-type metastatic colorectal cancer patients, who are BEAMing positive (KRAS mutated in blood) before treatment may have worse evolution in terms of PFS (progression Free Survival) and response rate than BEAMing negative (KRAS native in blood) patients.

To know the proportion of patients who are BEAMing positive (KRAS mutation can be detected in circulating extracellular DNA) at the beginning of treatment, could be of great importance for treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV colorectal adenocarcinoma.
* Patient ≥ 18 years of age.
* ECOG PS 0-1
* Life expectancy ≥ 6 months
* Candidate for first-line systemic chemotherapy according to regular clinical practice.
* Measurable disease.
* Wild-type KRAS
* Signed informed consent form.

Exclusion Criteria:

* Patient who has received prior chemotherapy for metastatic CRC, except for adjuvant treatment completed at least six months before entering study.
* Patient in whom there is a contraindication for the use of any of the drugs used in first-line treatment of colorectal cancer: 5-fluorouracil,, irinotecan or cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cáncer and wild-type KRAS treated with Folfiri-Cetuximab as first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the proportion of patients with advanced colorectal cancer in whom KRAS mutation can be detected in circulating extracellular DNA | Baseline

SECONDARY OUTCOMES:
To estimate the proportion of patients with metastatic colorectal cancer who switch from BEAMing negative to BEAMing positive while being treated with first line FOLFIRI-Cetuximab | At 4 months and every eight weeks until disease progression up to 12 months
To estimate the response rate, in biopsy-proven K-ras wild-type patients according to KRAS status in circulating extracellular DNA. | Every eight weeks until disease progression up to 12 months
Disease control rate according to KRAS status in circulating extracellular DNA. | Every eight weeks until disease progression up to 12 months
Complete response rate according to KRAS status in circulating extracellular DNA. | Every eight weeks until disease progression up to 12 months
Duration of response according to KRAS status in circulating extracellular DNA. | Every eight weeks until disease progression, up to 12 months
  From date of first documented response until de date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Early tumor shrinkage | At 4 months
Number of each adverse event per cycle | Every 2 weeks, until end of treatment, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, Doctor, Principal Investigator — Madrid Norte Sanchinarro University Hospital
Locations (1):
- Centro Integral Oncólógico Clara Campal (Madrid Norte Sanchinarro University Hospital), Madrid, Madrid, Spain